CLINICAL TRIAL: NCT02087540
Title: A Randomized, Double-blind, Multi-center, Factorial Phase III Clinical Trial to Evaluate the Efficacy and Safety of Telmisartan/Rosuvastatin Co-administration in Hypertensive Patients With Hyperlipidemia
Brief Title: Efficacy and Safety of Telmisartan/Rosuvastatin Co-administration in Hypertensive Patients With Hyperlipidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID_Telotan_1203
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Telmisartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Telmisartan 80mg & Rosuvastatin 20mg (Experimental): PO, Once Daily, 8 weeks
  Interventions: Drug: Telmisartan 80mg; Drug: Rosuvastatin 20mg; Drug: Placebo(for Rosuvastatin 10mg)
- Telmisartan 80mg & Rosuvastatin 10mg (Experimental): PO, Once Daily, 8weeks
  Interventions: Drug: Telmisartan 80mg; Drug: Rosuvastatin 10mg; Drug: Placebo(for Rosuvastatin 20mg)
- Telmisartan placebo & Rosuvastatin 20mg (Active Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Rosuvastatin 20mg; Drug: Placebo(for Telmisartan 80mg); Drug: Placebo(for Rosuvastatin 10mg)
- Telmisartan Placebo & Rosuvastatin 10mg (Active Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Rosuvastatin 10mg; Drug: Placebo(for Telmisartan 80mg); Drug: Placebo(for Rosuvastatin 20mg)
- Telmisartan 80mg & Rosuvastatin placebo (Active Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Telmisartan 80mg; Drug: Placebo(for Telmisartan 80mg); Drug: Placebo(for Rosuvastatin 20mg)
- Telmisartan placebo & Rosuvastatin placebo (Placebo Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Placebo(for Telmisartan 80mg); Drug: Placebo(for Rosuvastatin 20mg); Drug: Placebo(for Rosuvastatin 10mg)

INTERVENTIONS:
Drug: Telmisartan 80mg
  Arms: Telmisartan 80mg & Rosuvastatin 10mg; Telmisartan 80mg & Rosuvastatin 20mg; Telmisartan 80mg & Rosuvastatin placebo
Drug: Rosuvastatin 20mg
  Arms: Telmisartan 80mg & Rosuvastatin 20mg; Telmisartan placebo & Rosuvastatin 20mg
Drug: Rosuvastatin 10mg
  Arms: Telmisartan 80mg & Rosuvastatin 10mg; Telmisartan Placebo & Rosuvastatin 10mg
Drug: Placebo(for Telmisartan 80mg)
  Arms: Telmisartan 80mg & Rosuvastatin placebo; Telmisartan Placebo & Rosuvastatin 10mg; Telmisartan placebo & Rosuvastatin 20mg; Telmisartan placebo & Rosuvastatin placebo
Drug: Placebo(for Rosuvastatin 20mg)
  Arms: Telmisartan 80mg & Rosuvastatin 10mg; Telmisartan 80mg & Rosuvastatin placebo; Telmisartan Placebo & Rosuvastatin 10mg; Telmisartan placebo & Rosuvastatin placebo
Drug: Placebo(for Rosuvastatin 10mg)
  Arms: Telmisartan 80mg & Rosuvastatin 20mg; Telmisartan placebo & Rosuvastatin 20mg; Telmisartan placebo & Rosuvastatin placebo

SUMMARY:
To identify efficacy and safety of Telmisartan/Rosuvastatin co-administration in hyperlipidemia control in hypertensive patients with hyperlipidemia compared to each monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men and women >18 years of age
* Subject who has one of 3 conditions classifed by Cardiovascular Risk Factors, 10-Year Risk, Blood Pressure, LDL-C, Coronary Artery Disease and Equivalent

Exclusion Criteria:

* Female who are pregnant, breastfeeding, or of childbearing potential, unwilling to practice adequate contraception throughout the study,.
* Other exclusions applied

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
•Change in seated diastolicblood pressure at 8 weeks compared to the base value | at the 8 weeks
Change in LDL-Cat 8 weeks compared to the base value (% change) | at the 8 weeks

SECONDARY OUTCOMES:
Change in seateddiastolic blood pressure | at 2,4 8 weeks
Change in seated systolic blood pressure | at 2,4,8weeks
Rate of patients achieving a therapeutic purpose according to JNC VII Guideline [therapeutic purpose for blood pressure: < 140/90 mmHg (however, < 130/80 mmHg for Group III)] | at 2, 4 and 8 weeks
Change in LDL-Cat compared to the base value (% change) | 2, 4 and 8 weeks
Change in TC, TG, HDL-C and Apolipoprotein B compared to the base value (% change) | at 2, 4 and 8 weeks
Rate of patients achieving a therapeutic purpose according to NCEP ATP III Guideline therapeutic purpose for LDL-C- (Group I: < 160 mg/dL, Group II: < 130 mg/dL, Group III: < 100 mg/dL) | at 2, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Saint Mary's Hosiptal, Seoul, South Korea